CLINICAL TRIAL: NCT00231387
Title: Rosiglitazone and Plaque Study: A 12 Month Randomised, Double-blind, Placebo-controlled, Magnetic Resonance Imaging Study to Evaluate the Effect of Rosiglitazone on the Structure and Composition of Carotid Atherosclerotic Plaques in Subjects With Type 2 Diabetes Mellitus and Coexisting Vascular Disease or Hypertension
Brief Title: Rosiglitazone And Plaque Study for Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRL-049563/351
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Non-insulin-dependent Diabetes Mellitus
Keywords: diabetes rosiglitazone plaque
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone

INTERVENTIONS:
Drug: rosiglitazone

SUMMARY:
This is a phase IIIb, randomised, double blind, placebo controlled, study in patients with type 2 diabetes mellitus and coexisting vascular disease or hypertension. The total duration of the study will be approximately 60 weeks. The aim of this study is to examine the potential beneficial effects of rosiglitazone on carotid atheroma in patients with type 2 diabetes mellitus and coexisting vascular disease or hypertension. It is hypothesised that treatment with rosiglitazone will lead to an decrease in plaque size. In addition, it is hoped that rosiglitazone will have a positive effect on plaque composition and stability.

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes.
* Co-existing vascular disease.
* At least 6 months of statin or fibrate therapy.
* HbA1c <10% at screening and with at least one atheromatous plaque causing 10-95% narrowing of the internal carotid artery.

Exclusion criteria:

* Patients with >2 concomitant oral anti-hyperglycaemic agents within 3 months of screening.
* Previous exposure to a thiazolidinedione.
* History of chronic insulin use.
* Use of investigational drug within 30 days.
* Systolic blood pressure (bp) > 170 mmHg or diastolic bp >100 mmHg.
* Severe or unstable angina.
* History of: gangrene, TIA, stroke, hepatic disease, alcohol or drug abuse, surgery of the carotid arteries or claustrophobia.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-09 (Actual); Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
The effect of 52 wks oral treatment with rosiglitazone in comparison to placebo on change from baseline of the plaque total wall volume in the carotid artery, in patients with type 2 dm and vascular disease/hypertension, using cardiac mri. | 52 Weeks

SECONDARY OUTCOMES:
These include magnetic resonance endpoints related to plaque lipid content, volume, plaque size and fibrous cap thickness. Colour duplex measurements, laboratory assays for glycaemia and lipids.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Center, London, United Kingdom